CLINICAL TRIAL: NCT06003738
Title: A Comparative Study Between the Postoperative Analgesic Effect of Pericapsular Nerve Group Block (PENG) and Fascia Iliaca Compartment Block (FICB) in Total Hip Arthroplasty: a Prospective Randomized Clinical Trial
Brief Title: Comparing Postoperative Pain After Pericapsular Nerve Block and Fascia Iliaca Block in Total Hip Arthroplasty
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Diaaeldin Badr Aboelnile, Lecturer of Anesthesia, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FMASU MD76/2023
Record Dates: First submitted 2023-07-12; First posted 2023-08-22 (Actual); Last update posted 2023-08-23 (Actual); Status verified 2023-08

CONDITIONS: Anesthesia

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The fascia iliaca compartment block group (Active Comparator): The first group 34 patients
  Interventions: Procedure: fascia iliaca compartment block; Procedure: palcebo pericapsular nerve block
- The pericapsular nerve block group (Active Comparator): The second group 34 patients
  Interventions: Procedure: pericapsular nerve block; Procedure: palcebo fascia iliaca compartment block

INTERVENTIONS:
Procedure: fascia iliaca compartment block — Block will be performed using an ultrasound machine with a high-frequency linear probe covered with a sterile sheath and 100 mm needle.
  The patient will be positioned supine to perform the block, the skin is disinfected and the transducer positioned to identify the femoral artery and the iliopsoas muscle and fascia iliaca. The transducer is moved laterally until the sartorius muscle is identified. The in-plane technique will be used, and the tip of the needle will be inserted between the fascia iliaca and iliopsoas muscle. a syringe containing 15ml of 0.25% bupivacaine will be injected.
  Other Names: FICB
  Arms: The fascia iliaca compartment block group
Procedure: pericapsular nerve block — The block will be performed using the curvilinear low-frequency ultrasound probe to be placed over the line parallel to the inguinal ligament then It will be rotated 45◦ to identify the anterior inferior iliac spine, the iliopubic eminence, and the psoas tendon. A 22-gauge, 80 mm echogenic needle will be inserted in an in-plane approach to place the tip in the musculofascial plane between the pubic ramus posteriorly and the psoas tendon anteriorly a syringe containing 15ml of 0.25% bupivacaine will be injected .
  Other Names: PENG
  Arms: The pericapsular nerve block group
Procedure: palcebo fascia iliaca compartment block — Block will be performed using an ultrasound machine with a high-frequency linear probe covered with a sterile sheath and 100 mm needle.
  The patient will be positioned supine to perform the block, the skin is disinfected and the transducer positioned to identify the femoral artery and the iliopsoas muscle and fascia iliaca. The transducer is moved laterally until the sartorius muscle is identified. The in-plane technique will be used, and the tip of the needle will be inserted between the fascia iliaca and iliopsoas muscle. a syringe containing 15ml of normal saline will be injected.
  Other Names: palcebo FICB
  Arms: The pericapsular nerve block group
Procedure: palcebo pericapsular nerve block — The block will be performed using the curvilinear low-frequency ultrasound probe to be placed over the line parallel to the inguinal ligament then It will be rotated 45◦ to identify the anterior inferior iliac spine, the iliopubic eminence, and the psoas tendon. A 22-gauge, 80 mm echogenic needle will be inserted in an in-plane approach to place the tip in the musculofascial plane between the pubic ramus posteriorly and the psoas tendon anteriorly a syringe containing 15ml of normal saline will be injected .
  Other Names: palcebo PENG
  Arms: The fascia iliaca compartment block group

SUMMARY:
The aim of this study is to investigate the efficiency of post-operative analgesia by fascia iliaca compartment block versus pericapsular nerve group block block in reducing narcotic consumption during the first 24 hour post-operatively by using the Visual Analogue Scale.

DETAILED DESCRIPTION:
Total hip arthroplasty is a widely used surgical treatment intervention for treating hip conditions such as femur neck fractures and advanced hip osteoarthritis.

Hip fractures are quite common, regardless of the age of the population (young or old), and they are extremely painful. A hip fracture is a serious injury with potentially life-threatening complications, and it is a common orthopedic emergency in elderly individuals. Early surgery within 48 hours of a fracture has been found to lower mortality and complication rates.

The pericapsular nerve group block is a novel regional analgesia technique to decrease pain after THA while preserving the motor function. The local anaesthetic is deposited using this method in the fascial plane between the psoas muscle and the superior pubic ramus, which aims sensory branches of the obturator, accessory obturator, and femoral nerves in the anterior capsule of the hip.

Fascia iliaca compartment block, for procedures on the femur and hip joint, is still a well-liked regional anaesthetic technique. Studies have found that FICB prevents complications by anaesthetizing the femoral nerve far from critical neurovascular structures while still giving enough analgesia.

Both blocks could be used to effectively reduce pain intensity up to 24 hours, total opioid consumption, and length of hospital stay in THA patients.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-80 years.
2. Sex: Both sexes.
3. American Society of Anaesthesiologists (ASA) Physical Status Class I, II, and III.
4. Scheduled for Total hip arthroplasty (THA) under spinal anesthesia.

Exclusion Criteria:

1. Declining to give a written informed consent.
2. History of allergy to the medications used in the study.
3. Contraindications to regional anesthesia (including patient refusal, coagulopathy, and local infection).
4. Psychiatric disorders.
5. Significant cognitive dysfunction.
6. American Society of Anesthesiologists (ASA) Physical Status Class IV.
7. Liver failure, renal insufficiency (estimated glomerular filtration rate < 15 mL/min/1.73 m2).
8. Patients who had failed spinal anaesthesia were excluded from the study.
9. Pregnancy.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Estimated)
Dates: Start 2023-08-21 (Actual); Primary Completion 2024-08-21 (Estimated); Study Completion 2024-09-01 (Estimated)

PRIMARY OUTCOMES:
The effect of the studied blocks on the Visual Analogue Scale for pain | Immediately postoperatively (zero time)
  the Visual Analogue Scale for pain is ranging from 0 to 10, where 0 is no pain and 10 is maximum pain
Change in the Visual Analogue Scale for pain | Every 2 hours during the first 6 hours
  the Visual Analogue Scale for pain is ranging from 0 to 10, where 0 is no pain and 10 is maximum pain
Change in the Visual Analogue Scale for pain | every 6 hours in the first 24 hours postoperatively
  the Visual Analogue Scale for pain is ranging from 0 to 10, where 0 is no pain and 10 is maximum pain

SECONDARY OUTCOMES:
The total dose of nalbuphine in mg was used postoperatively per patient | 24 hours postoperatively
  rescue analgesia
Mean arterial blood pressure change | 24 hours postoperatively
  hemodynamics
Heart rate change | 24 hours postoperatively
  hemodynamics

CONTACTS AND LOCATIONS:
Overall Officials: Diaaeldin DA Aboelnile, MD, Lecturer, Principal Investigator — Faculty of Medicine, Ain Shams University
Locations (1):
- Ain shams university hospitals, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No